CLINICAL TRIAL: NCT00796107
Title: An Open Label Study to Evaluate the Safety, Tolerability and Effect on Tumor Response of R1507 in Combination With Letrozole in Postmenopausal Women With Advanced Breast Cancer.
Brief Title: A Study of R1507 in Combination With Letrozole in Postmenopausal Women With Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the discontinuation of compound development, this study has been terminated.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO21161
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — RG-1507 monoclonal antibody; Letrozole

ARMS (1):
- R1507 in Combination With Letrozole (Experimental): Participants received a full daily dose of 2.5 mg of orally administered Letrozole along with 16 mg/kg of intravenous R1507 administered q3w, and observed for dose limiting toxicity for the first 2 cycles of treatment.
  Interventions: Drug: RG1507; Drug: Letrozole

INTERVENTIONS:
Drug: RG1507 — R1507 was administered at a dose 16 mg/kg every 3 weeks.
Drug: Letrozole — Letrozole was administered orally at a dose 2.5 mg daily.

SUMMARY:
This study aim was to determine the safety and efficacy of R1507 in combination with letrozole in patients with advanced breast cancer. In the first part of the study a cohort of patients with advanced breast cancer received letrozole 2.5mg po daily in combination with R1507 16mg/kg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal female patients;
* stage IV or locally advanced breast cancer;
* measurable disease;
* letrozole failure (Part 2);
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.

Exclusion Criteria:

* previous chemotherapy for metastatic breast cancer;
* concurrent antibody or immunotherapy for advanced disease, within 4 weeks prior to receipt of study drug;
* history of primary malignancy in 5 years prior to study, excluding adequately treated basal or squamous cell cancer of skin, or cancer in situ of cervix;
* concurrent radiotherapy, or radiotherapy within 28 days prior to receipt of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01-28 (Actual); Primary Completion 2010-03-03 (Actual); Study Completion 2010-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Atlanta, Georgia
  - St Louis, Missouri
  - Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R1507 in Combination With Letrozole
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 1
Not completed — Progressive Disease | 5

BASELINE CHARACTERISTICS:
Arm/Group | R1507 in Combination With Letrozole
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Part 2)
Time Frame: Up to 14 months
Population: Phase 2 of this study was not conducted.
Arm/Group | R1507 in Combination With Letrozole
Number analyzed (Participants) | 0

2. Secondary Outcome: Pharmacokinetics (PK) Profile (Part 2)
Time Frame: Up to 14 months
Population: Phase 2 of this study was not conducted.
Arm/Group | R1507 in Combination With Letrozole
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival (Part 2)
Time Frame: Up to 14 months
Population: Phase 2 of this study was not conducted.
Arm/Group | R1507 in Combination With Letrozole
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Adverse Events (Part 2)
Time Frame: Up to 14 months
Population: Since Phase 2 of this study was not conducted, this outcome measure was not collected.
Arm/Group | R1507 in Combination With Letrozole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 13 months
Arm/Group | R1507 in Combination With Letrozole
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R1507 in Combination With Letrozole (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R1507 in Combination With Letrozole (N=6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Blood creatinine increased (Investigations) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diastolic Dysfunction (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Irritability (General disorders) | 1 (1)
Oral Candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Decreased Apetite (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Phase 2 of this study was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.